CLINICAL TRIAL: NCT01426321
Title: Individually Tailored Cardiac Resynchronization Therapy - Combing Myocardial Strain and Cardiac CT to Optimize Left Ventricular Lead Placement in Cardiac Resynchronization Therapy
Brief Title: Combining Myocardial Strain and Cardiac CT to Optimize Left Ventricular Lead Placement in CRT Treatment
Acronym: CRT clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Crafoord Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRTCLIN01
Record Dates: First submitted 2011-08-25; First posted 2011-08-31 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronization therapy; Echocardiography; Cardiac computed tomography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imaging guided LV lead positioning (Active Comparator)
  Interventions: Other: Imaging guided LV lead positioning
- Standard LV lead positioning (No Intervention): The LV lead position is decided at the discretion of the treating physician. Cardiac CT images are available for viewing, but no echocardiography data regarding segmental myocardial strain are available.

INTERVENTIONS:
Other: Imaging guided LV lead positioning — LV lead positioning guided by echocardiography (mechanical strain evaluation by speckle tracking) in combination with cardiac CT. A viable segment with the latest mechanical activation is targeted, and an appropriate "optimal" cardiac vein segment is then chosen using the CT images.
  Arms: Imaging guided LV lead positioning

SUMMARY:
For patients with advanced heart failure, Cardiac Resynchronization Therapy (CRT) has been a major improvement. The treatment improves symptoms and prolongs life in selected patients with heart failure. However, with the current selection criteria and methods for implanting the pacemaker, only 60-70% of the patients derive significant benefit from the treatment.

New imaging techniques, including advanced ultrasound and computed tomography, in combination with new versatile multi-pole electrodes, have made an individually tailored therapy possible. Using these techniques in combination, the study will investigate the effect of individually based "optimal" placement of the pacemaker electrodes vs. standard care. The optimal LV electrode position is defined as pacing a viable segment with the latest mechanical delay, targeting a specific segment of the coronary sinus as visualised on cardiac CT. The hypothesis is that this will increase the number of positive responders from 65% to 85%.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure (New York Heart Association functional class II - IV) despite stabile optimal medical therapy.
* Wide QRS ≥ 120 milliseconds on standard ECG.
* LV systolic dysfunction (EF ≤ 35%).
* Written informed consent.
* Accepted for CRT-P or CRT-D treatment

Exclusion Criteria:

* Life expectancy < 12 months.
* Recent myocardial infarction (< 3 months).
* Significant valve disease
* Chronic atrial fibrillation
* Pregnancy
* Severely impaired renal function (estimated glomerular filtration rate (eGFR) < 30 ml/min)
* Unable to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Positive response to CRT treatment | 6 months
  The primary efficacy endpoint will evaluate the effect of echocardiography and cardiac CT guided placement of the left ventricular lead vs standard care (i.e. position of the left ventricular lead at the discretion of the treating physician).
  Number of patients with positive response to CRT (YES or NO). A positive response is defined as survival in combination with either a reduction in end systolic left ventricular volume ≥ 15% by echocardiography ("volume responder") and / or improvement ≥ 1 NYHA class and ≥10% improvement in 6 minute hall walk test ("clinical responder").

SECONDARY OUTCOMES:
Response to CRT (on-treatment analysis) | 6 months
  Evaluate the effect of optimal LV placement (post hoc analysis of both groups) versus non-optimal LV lead placement. Optimal lead placement is defined as pacing from a viable segment with the latest mechanical activation (by myocardial strain measurement). Outcome measure is the same as in the primary outcome measure.
Heart failure morbidity | 6 months 2 years and 5 years
  Evaluate the effect of echocardiography guided LV lead placement compared to standard care in relation to hospitalisation for worsening of heart failure
Morbidity and mortality | 6 months 2 years and 5 years
  Evaluate the effect of echocardiography guided LV lead placement compared to standard care in relation to a composite endpoint of all cause mortality and hospitalisation for worsening of heart failure (2 years and 5 years).
Mortality | 6 months, 2 years and 5 years
  Evaluate the effect of echocardiography guided LV lead placement compared to standard care in relation to all cause mortality
Left ventricular dyssynchrony | 6 months
  Evaluate the effect of echocardiography guided LV lead placement compared to standard care in relation to echocardiography measured changes in LV dyssynchrony
Ventricular tachycardia | 6 months 2 years and 5 years
  Evaluate the effect of echocardiography guided LV lead placement compared to standard care in relation to number of treated ventricular tachycardia episodes
Quality of life | 6 months 2 years 5 years
  Evaluate the effect of echocardiography guided LV lead placement compared to standard care in relation to the change in the Minnesota Living with heart failure Quality of Life questionnaire
Myocardial viability | Peroperative
  Evaluate the concordance in viability assessment using myocardial strain evaluation (echocardiography) compared to cardiac MRI.
Biochemical markers of heart failure | 6 months
  Evaluate the effect of echocardiography guided LV lead placement compared to standard care in relation to the change in blood natriuretic peptide (BNP) levels
Left ventricular systolic function | 6 months
  Evaluate the effect of echocardiography guided LV lead placement compared to standard care in relation to the change in LV ejection fraction
Myocardial viability | 6 months
  Evaluate the concordance between echocardiography (strain evaluation with speckle tracking) and cardiac MRI viability images (late gadolinium enhancement).
MRI left ventricular dyssynchrony | 6 months
  Evaluate if MRI dyssynchroni evaluation has incremental value over echocardiography alone for predicting the effect of cardiac resynchronization therapy.
Left ventricular diastolic dimension | 6 months
  Evaluate the effect of echocardiography guided LV lead placement compared to standard care in relation to the change in left ventricular diastolic dimension

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Borgquist, MD PhD, Principal Investigator — Region Skane
Locations (1):
- Skane University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Borgquist R, Carlsson M, Markstad H, Werther-Evaldsson A, Ostenfeld E, Roijer A, Bakos Z. Cardiac Resynchronization Therapy Guided by Echocardiography, MRI, and CT Imaging: A Randomized Controlled Study. JACC Clin Electrophysiol. 2020 Oct;6(10):1300-1309. doi: 10.1016/j.jacep.2020.05.011. Epub 2020 Aug 12. PMID 33092758